CLINICAL TRIAL: NCT05723081
Title: The Impact of Structural Racism and Discrimination (SRD) on Mechanisms of the Native American Pain Disparity
Brief Title: Oklahoma Study of Native American Pain Risk III: Stress and Resilience
Acronym: OK-SNAPIII
Status: Recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma State University (Other); University of Tulsa (Other)
Responsible Party: Sponsor
Other Study IDs: HSC16494/TU2229
Record Dates: First submitted 2023-01-24; First posted 2023-02-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Discrimination, Racial; Stress Physiology; Pain
Keywords: Structural racism and discrimination; Stress reactivity; Quantitative sensory testing
MeSH Terms: conditions — Racism; Pain; Systemic Racism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Participants will provide 20 saliva samples during the study to measure salivary cortisol. Participants will also provide small samples of blood via finger stick to assess glucose regulation (HbA1c), systemic inflammation (hs-CRP), and a lipid profile (i.e., HDL, LDL, triglycerides, cholesterol.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Native Americans: Native Americans / American Indians

SUMMARY:
The goal of this observational study is to learn about the relationship between environmental structural racism and discrimination and chronic pain risk in Native American adults. The main questions it aims to answer are:

1. How does environmental structural racism and discrimination affect chronic pain-promoting mechanisms in Native Americans?
2. What psychosocial factors buffer the negative effects of environmental structural racism and discrimination on chronic pain-promoting mechanisms?

DETAILED DESCRIPTION:
Native Americans experience higher rates of chronic pain than the general U.S. population, and previous research has shown that pain-free Native Americans transition to chronic pain at almost three times the rate of non-Hispanic Whites. Yet, little is known about the mechanisms that contribute to this pain disparity.

This study aims to better understand the role of environmental and society-wide stressors, like structural racism and discrimination, in contributing to this pain disparity. It is believed that these environmental and social stressors may contribute to chronic pain risk by increasing an individual's mental and physical stress levels. In turn, increased stress may alter how an individual responds to pain, both physically and emotionally, which may place them at greater risk for developing chronic pain in the future.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Native American/American Indian

Exclusion Criteria:

* <18 years of age
* Self-reported history of cardiovascular, neuroendocrine, musculoskeletal, or neurological disorders
* Surrent chronic pain, defined as persistent, bothersome pain on more days than not for at least 3 months)
* Self-reported current substance dependence
* Sse of medication that could interfere with testing (e.g., recent use of analgesics, antidepressants, or anti-anxiety medications)
* Inability to speak English
* Current psychosis (assessed by Psychosis Screening Questionnaire)
* Serious cognitive impairment (assessed by <20 score on the Montreal Cognitive Assessment [MoCA])
* Possible peripheral neuropathy (assessed by nerve conduction study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be adults who self-identify as Native American/American Indian.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain inhibition | baseline
  Pain inhibition will be assessed using a conditioned pain modulation task with cold water as the conditioning stimulus and electric stimulations as the test stimulus.
Inhibition of pain-related spinal reflex | baseline
  Pain-related spinal reflex inhibition assessed from electromyogram will be assessed using a conditioned pain modulation task with cold water as the conditioning stimulus and electric stimulations as the test stimulus.
Inhibition of pain-evoked cortical potentials | baseline
  Inhibition of pain-evoked cortical potentials from electroencephalography will be assessed using a conditioned pain modulation task with cold water as the conditioning stimulus and electric stimulations as the test stimulus.
Psychological stress | baseline
  A single latent variable measuring psychological stress will be created using principal components analysis to combine scores from three self-report questionnaires: the Perceived Stress Scale (PSS), the Global Distress Index of the Symptom Checklist-90-Revised (SCL-90-R), and the PTSD Checklist-Civilian (PCL-C).
Somatic threat sensitivity | baseline
  A single latent variable measuring somatic threat sensitivity will be created using principal components analysis to combine scores from the Pain Catastrophizing Scale and a pain-related anxiety visual analog scale.
Allostatic load | baseline
  A single latent variable for allostatic load will be created using principal components analysis to combine cardiovascular (i.e., resting blood pressure and heart rate, stress-evoked blood pressure and heart rate, and a fasting lipids profile [HDL, LDL total cholesterol, and triglycerides]), metabolic (i.e., BMI, waist-to-hip ratio, HbA1c), neuroendocrine (i.e., diurnal salivary cortisol, stress-evoked salivary cortisol), immune (i.e., hs-CRP), and parasympathetic (i.e., resting heart rate variability) variables.
Environmental structural racism and discrimination | baseline
  An index comprised of 11 environmental justice variables from the Environmental Protection Agency's publicly available Environmental Screening and Mapping Tool (EJSCREEN) will be created for each participant at the 2010 Census Block Group level. The 11 variables will be combined into a single index using principal components analysis.
Cultural connectedness | baseline
  A single latent variable of cultural connectedness will be created using principal components analysis to combine scores from five self-report scales: the Cultural Connectedness Scale, the Community Mastery Scale, the Vancouver Index of Acculturation, the American Indian Enculturation Scale, and the Native American Spirituality Scale

SECONDARY OUTCOMES:
Temporal summation of pain | baseline
  Temporal summation of pain will be measured by assessing the change in a participant's pain ratings in response identical noxious stimuli delivered in rapid succession.
Temporal summation of spinal nociception | baseline
  Temporal summation of spinal nociception will be measured by assessing the change in a participant's pain-related reflex magnitude (assessed from electromyography) in response identical noxious stimuli delivered in rapid succession.
Pain tolerance | basline
  Pain tolerance will be measured with ischemic and cold pain tasks. Participants will continuously rate their pain in response to painful tonic stimuli, and pain tolerance will be quantified as the time (in seconds) that it takes for participants to report that they can no longer tolerate the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Rhudy, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma - Schusterman Center, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Immediately following publication of all findings, the data will be freely available to any researcher who requests a copy. All data files will be de-identified so there is no possibility of connecting the information with the original participants. The electronic data will be stored as de-identified SPSS data files or Excel data files. The raw (i.e., unprocessed) physiology data (e.g., EMG, EKG, EEG) will also be made available to interested researchers. These raw data files will be stored as de-identified files. To obtain access to the data, interested parties can contact the PI (jamie-rhudy@utulsa.edu).
Time Frame: De-identified data will become available following publication of all findings (around 6/1/2030).
Access Criteria: To obtain access to the data, interested parties can contact the PI (jamie-rhudy@utulsa.edu).